CLINICAL TRIAL: NCT04195360
Title: Postoperative Incidence of Orthostatic Intolerance and Hypotension in Patients Undergoing Primary Unicompartmental Knee Arthroplasty (UKA)
Brief Title: Postoperative Incidence of Orthostatic Intolerance and Hypotension in Primary Unicompartmental Knee Arthroplasty (UKA)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Kehlet, Henrik, M.D., Ph.D. (Individual)
Responsible Party: Principal Investigator, Louise Bundsgaard Andersen, Undergraduate Student, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-19063289
Record Dates: First submitted 2019-12-02; First posted 2019-12-11 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Orthostatic Hypotension; Orthostatic Intolerance; Postoperative Complications
MeSH Terms: conditions — Hypotension, Orthostatic; Orthostatic Intolerance; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Orthostatic intolerant (OI): Patients that experience symptoms of orthostatic intolerance (dizziness, nausea, vomiting, blurry vision or syncope) or orthostatic hypotension (fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg) during mobilization
  Interventions: Other: Standardized mobilization procedure
- Orthostatic tolerant (OT): Patients that do not experience symptoms of orthostatic intolerance (dizziness, nausea, vomiting, blurry vision or syncope) or orthostatic hypotension (fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg) during mobilization
  Interventions: Other: Standardized mobilization procedure

INTERVENTIONS:
Other: Standardized mobilization procedure — 5 minutes bed rest (h1), followed by 3 minutes passive leg raise (PLR), followed by 5 minutes bed rest (h2), followed by 3 minutes sitting on the egde of the bed (sit), followed by 3 minutes standing/walking on the spot (sta), followed by 5 minutes bedrest (h3)

SUMMARY:
Incidence and pathophysiologic hemodynamics of orthostatic intolerance and orthostatic hypotension in patients undergoing UKA

DETAILED DESCRIPTION:
In today's multimodal fast-track perioperative care program (ERAS) early mobilization is an essential cornerstone, and is known to prevent postoperative morbidity and lower length of stay in the hospital. Intact orthostatic blood pressure regulation is necessary to complete mobilization, and postoperative orthostatic hypotension (OH), defined as a drop in systolic arterial pressure (SAP) > 20 mmHg or a drop >10 mmHg in diastolic arterial pressure (DAP) and orthostatic intolerance (OI), characterized by dizziness, nausea, feeling warm and syncope related to orthostatic challenge, are well-known reasons for delayed early mobilization, prolonged bedrest and delayed ambulation.

Former studies have been accessing the postoperative incidence in THA-patients (22%-40%), TKA-patients(36%), colorectal patients(53%), abdominal and cardiothoracic surgery patients(40%), radical prostatectomy patients (50%). One study have been accessing the postoperative incidence of OI in mastectomy patients and found an incidence of 4%, and thereby indicating that postoperative OI is not an issue in minor surgery.

This study is the first, to our acknowledgement, which accesses the postoperative incidence of OI/OH in UKA-patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and
* Patients undergoing UKA in spinal anesthesia at Hvidovre Hospital in a standardized fast-track setting.
* Patients that speak and understand Danish
* Written informed consent

Exclusion Criteria:

* Pre-existing orthostatic hypotension or intolerance
* Alcohol or substance abuse
* everyday treatment with either anxiolytic or antipsychotic medicine
* Cognitive dysfunction
* If surgery was converted to general anesthesia or total knee arthroplasty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were screened in the electronic patient system, and were first screened for inclusion criteria, and afterwards exclusion criteria.
  Patients were eligible to enroll in the study if they were >18 years, spoke and understood Danish, signed an informed consent formula and underwent UKA in spinal anesthesia at Hvidovre Hospital. They were excluded if they had 1) pre-existing orthostatic hypotension or intolerance, 2) Alcohol or substance abuse, 3) everyday treatment with either anxiolytic or antipsychotic medicine 4) Cognitive dysfunction. 5) Or if surgery was converted to general anesthesia or total knee arthroplasty.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of orthostatic intolerance | 6 hours postoperatively
  Symptoms of orthostatic intolerance: dizziness, nausea, vomiting, blurry vision or syncope during mobilization
Incidence of orthostatic hypotension | 6 hours postoperatively
  Orthostatic hypotension is defined as a fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg during mobilization

SECONDARY OUTCOMES:
Changes in systolic arterial pressure (SAP) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg, LiDCO-apparatus
Changes in diastolic arterial pressure (DAP) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg, LiDCO-apparatus
Changes in mean arterial pressure (MAP) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg, LiDCO-apparatus
Changes in cardiac output (CO) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL/min, LiDCO-apparatus
Changes in systemic vascular resistance (SVR) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg⋅min⋅mL-1
Changes in stroke volume (SV) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL, LiDCO-apparatus
Changes in heart rate variability (HRV) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in ms, LiDCO-apparatus
Changes in peripheral perfusion index (PPI) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in arbitrary units (AU), Massimo apparatus
Changes in cerebral perfusion (ScO2) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in %, NIRS-apparatus
Changes in muscular perfusion (SmO2) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in %, NIRS-apparatus
Changes in haemoglobin (Hgb) concentration | Preoperatively, 6 and 24 hours postoperatively
  Measured in millimoles/L
Changes in C-Reactive Protein | Preoperatively, 6 and 24 hours postoperatively
  Measured in mg/L

OTHER OUTCOMES:
Pain score during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured by verbal rating scale (VRS) from 0 to 10
Estimated bleeding | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL
Opioid usage | Preoperatively, 6 and 24 hours postoperatively
  Measured in mg
Cumulative fluid administration and losses | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hristovska AM, Andersen LB, Uldall-Hansen B, Kehlet H, Troelsen A, Gromov K, Foss NB. Postoperative orthostatic intolerance following fast-track unicompartmental knee arthroplasty: incidence and hemodynamics-a prospective observational cohort study. J Orthop Surg Res. 2024 Apr 1;19(1):214. doi: 10.1186/s13018-024-04639-6. PMID 38561817